CLINICAL TRIAL: NCT06041568
Title: A Phase 1b, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Imvotamab in Participants With Severe Systemic Lupus Erythematosus Who Have Failed Standard Therapies
Brief Title: A Study of Imvotamab in Severe Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Decision.
Sponsor: IGM Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGM-2323-101
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Systemic Lupus Erythematosus; Lupus Erythematosus
Keywords: Lupus; SLE; Severe Lupus; Severe systemic lupus erythematosus; Systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imvotamab (Dose Escalation) (Experimental): Imvotamab administered intravenously
  Interventions: Drug: Imvotamab

INTERVENTIONS:
Drug: Imvotamab — Administered intravenously

SUMMARY:
The purpose of this study is to determine the safety and tolerability of imvotamab in patients with severe systemic lupus erythematosus who have failed prior therapies.

Participants will be given imvotamab through a vein (i.e., intravenously).

DETAILED DESCRIPTION:
This is a Phase 1b, randomized, placebo-controlled, multicenter study to determine the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of imvotamab in adult participants with systemic lupus erythematosus (SLE). Approximately 18 participants will be assigned to different sequentially dose escalation cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years at the time of signing ICF
* Diagnosis of SLE according to the 2019 European League Against Rheumatism/American College of Rheumatology (ACR) Classification Criteria at least 16 weeks or more prior to screening
* Highly active SLE disease, as demonstrated by a total systemic lupus erythematosus disease activity index (SLEDAI-2K) total score of ≥ 10 at screening
* Active SLE disease despite treatment with at least 1 immunosuppressive or biologic standard-of-care agent (e.g., methotrexate, azathioprine, mycophenolate mofetil, belimumab, anifrolumab) determined at the discretion of the investigator after at least 3 months of treatment.
* It must be planned that the background standard-of-care treatment remains at a stable dose throughout the Screening Period and up to Week 8.

Key Exclusion Criteria:

* Pregnant or breastfeeding or intending to become pregnant during the study or within 3 months after the final dose of imvotamab.
* Any lupus-associated neuropsychiatric disease.
* Active lupus nephritis with estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2, calculated according to the Chronic Kidney Disease Epidemiology Collaboration equation, classified as World Health Organization (WHO) Class IV.
* Prednisone-equivalent > 30 mg/day, including immediate and extended-release oral formulations.
* Drug-induced lupus.
* Participants with a history of catastrophic or severe anti-phospholipid syndrome within 12 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of imvotamab | Up to Week 52
  Incidence of adverse events (AEs), serious adverse events (SAEs), including serious infectious events and opportunistic infections

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kunder, Study Director — IGM Biosciences
Locations (10):
- United States (8):
  - TriWest Research Associates, San Diego, California
  - East Bay Rheumatology, San Leandro, California
  - Omega Research, DeBary, DeBary, Florida
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - Stryde Research, Allen, Texas
  - Precision Comprehensive Clinical Research, Grapevine, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Care and Cure Clinic, Houston, Texas
- Niepubliczny Zakład Opieki Zdrowotnej Lecznica MAK-MED w Nadarzynie, Nadarzyn, Poland
- Seoul National University Hospital, Seoul, South Korea